CLINICAL TRIAL: NCT05456074
Title: Integrative Molecular Characterization Of MiT Family Translocation Renal Cell Carcinomas (IMCOR)
Acronym: IMCOR
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Institut de cancérologie Strasbourg Europe (Other)
Collaborators: National Cancer Institute, France (Other Government); Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: 4-2021-001
Record Dates: First submitted 2022-07-08; First posted 2022-07-13 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Renal Carcinoma
Keywords: MiT family translocation renal cell carcinomas; Multiomics; Genetic; Epigenetic
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Tumor samples (DNA and RNA extraction)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with TRCC
  Interventions: Other: Data collection
- Patients with other rare kidney tumors
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection — Retrospective data collection

SUMMARY:
Microphthalmia transcription factor (MiT) family translocation renal cell carcinomas (TRCC) are rare subtypes of kidney cancers, which often arise in children and young adults. TRCC are characterized by translocations affecting transcription factors: Transcription Factor Binding To Immunoglobulin Heavy Constant Mu Enhancer 3 (TFE3) and Transcription Factor EB (TFEB). Little is known about TRCC molecular heterogeneity, in particular their transcriptomic and epigenetic subtype classification. Clinical behavior of TRCC is varying with age and Tumor, Node, Metastasis (TNM) stage. However, the biological basis of this aggressiveness is poorly understood.

PURPOSE: The primary goal of this study is to decipher specific alterations in aggressive TRCC, defined as cases with metastatic dissemination at diagnosis. To tackle this problem, a retrospective cohort of TRCC cases in children and young adults will be created. We will then perform integrative comprehensive multi-omics analysis of these tumors to identify genetic, epigenetic and immune biomarkers associated with metastatic behavior in a training and validation datasets. Comparison of the multi-omics data will be compared to other type of rare Kidney tumors as well as clear-cell renal cell carcinomas

DETAILED DESCRIPTION:
This retrospective cohort study aims to allow tumor collection of TRCC from three different networks: the French research network in renal cancer (UroCCR), the International Society of Paediatric Oncology (SIOP) database and the network for rare renal carcinomas (CARARE). Those samples will be divided in training and validation datasets. We will also collect samples from patients with other rare kidney cancers and clear-cell renal cell carcinomas allowing comparisons of similarity and differences between these tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients treated for kidney cancer in a clinical center located in France

For molecular biology study :

* Patients with tumor sample available for genetic and epigenetic analysis. Tumor sample stored in Biological resource facilities and consent given from patient or from parents for the use of biological sample for biomedical research purposes.

Exclusion Criteria:

* Objection from patient or parents

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with TRCC and other rare kidney tumors
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-01-25 (Estimated); Primary Completion 2026-01-25 (Estimated); Study Completion 2026-01-25 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic alterations associated with TRCC aggressiveness. | at the end of the study (36 months)
  Tumor aggressiveness is defined as TRCC cases with metastatic dissemination at diagnosis. Comparison of recurrent genetic aberration identified between metastatic and localized cases.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From renal tumor diagnosis to progression or latest patient news at the end of the study (36 months)
  Testing for association between molecular tumor features and clinico-pathological patients outcome, PFS, according to the identity of TFE fusion partner
Overall survival (OS) | From renal tumor diagnosis to death or latest patient news at the end of the study (36 months)6 months)
  Testing for association between molecular tumor features and clinico-pathological patients outcome, OS, according to the identity of TFE fusion partner
Contribution of DNA methylation, transcriptome and immune landscape to metastatic potential | at the end of the study (36 months)
  Proportion of patients with metastatic disease in each DNA methylation and messenger RNA (mRNA) cluster using hierarchical unsupervised subtype classifications

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel MALOUF, MD, PhD, Principal Investigator — Institut de cancérologie Strasbourg Europe
Locations (4):
- France (4):
  - Réseau Français de Recherche sur le Cancer du Rein (UroCCR), Bordeaux
  - Réseau SIOP, Hôpital Trousseau, Paris
  - Réseau CARARE, Rennes
  - Institut de cancérologie Strasbourg Europe, Strasbourg

REFERENCES:
- [Background] Herrscher H, Boileve A, Lindner V, Barthelemy P, Hutt E, Pierard L, Kurtz JE, Rioux-Leclercq N, Lang H, Malouf GG. [MiT family translocation renal cell carcinomas: Natural history, molecular features and multidisciplinary management]. Bull Cancer. 2020 Feb;107(2):272-280. doi: 10.1016/j.bulcan.2019.11.010. Epub 2020 Feb 7. French. PMID 32044098